CLINICAL TRIAL: NCT00455026
Title: Effect of Remifentanil on Electroencephalographic BAR Index During Propofol Anaesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Biopharmica Limited (Industry)
Responsible Party: David Breeze, Cortical Dynamics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2005.236
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-03

CONDITIONS: Depth of Anaesthesia
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): 0 ng/ml target effect site concentration remifentanil
  Interventions: Drug: remifentanil
- 2 (Active Comparator): 2 ng/ml target concentration remifentanil
  Interventions: Drug: remifentanil
- 3 (Active Comparator): 4 ng/ml target effect site concentration remifentanil
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — target effect site concentration during induction
  Other Names: No other names

SUMMARY:
Current cortical EEG based depth of anaesthesia monitors do not accurately reflect the effect of opioid drugs. We have developed a new theoretically-based method of analysing the EEG. Our hypothesis is that this new method will more accurately predict depth of anaesthesia than the Bispectral Index (BIS) monitor in patients having elective surgery.

DETAILED DESCRIPTION:
Patients aged 18-60 years presenting for elective surgery under general anaesthesia will be recruited. They will be randomised to receive remifentanil effect-site target 0, 2 or 4 ng/ml. Then anaesthesia will be induced with propofol. Loss of the eyelash reflex, response to command and response to electrical stimulation will be measured. The raw EEG will be recorded and analysed off-line using our new method and also for BIS values. Anaesthesia will then proceed according to the needs of the patient and the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18-60 years, of ASA physical status 1-3, presenting for elective surgery under general anaesthesia

Exclusion Criteria:

* Inadequate English comprehension due to a language barrier, cognitive deficit or intellectual disability
* Epilepsy or other EEG abnormality
* Prescription or illicit drugs known to affect the EEG

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Prediction probability for prediction of anaesthetic endpoints | During induction of anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (2):
- Australia (2):
  - Swinburne University, Hawthorn, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria